CLINICAL TRIAL: NCT06133634
Title: Clinical Translation of Senolytic Therapy With Fisetin to Improve Vascular Function in Older Adults
Brief Title: Fisetin to Improve Vascular Function in Older Adults
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Colorado, Boulder (Other)
Collaborators: American Heart Association (Other)
Responsible Party: Principal Investigator, Matthew Rossman, Assistant Research Professor, University of Colorado, Boulder
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 23-0288
Record Dates: First submitted 2023-11-10; First posted 2023-11-15 (Actual); Last update posted 2025-11-12 (Actual); Status verified 2025-11

CONDITIONS: Aging; Endothelial Dysfunction; Arterial Stiffness
MeSH Terms: interventions — fisetin

STUDY DESIGN:
Intervention Model Description: Randomized, double-blind, placebo-controlled, parallel group design clinical trial.
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fisetin (Active Comparator): Fisetin will be administered in an intermittent manner with two, three-day dosing periods at a dose of 2 mg/kg/day separated by two weeks.
  Interventions: Dietary Supplement: Fisetin
- Placebo (Placebo Comparator): Placebo capsules identical in appearance to fistin capsules will be administered in an intermittent manner with two, three-day dosing periods separated by two weeks.
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Fisetin — Fisetin dietary supplement
  Arms: Fisetin
Other: Placebo — Placebo capsules identical in appearance to fisetin capsules
  Arms: Placebo

SUMMARY:
This is a pilot clinical trial to test the efficacy of intermittent treatment with the flavonoid compound fisetin for improving vascular endothelial function and reducing aortic stiffness in older adults. This trial will also determine the potential mechanisms by which fisetin may improve vascular function, including by decreasing mitochondrial oxidative stress, cellular senescence and senescence-associated secretory phenotype (SASP) factors in circulation. Lastly, safety, tolerability and adherence of fisetin treatment will be assessed.

DETAILED DESCRIPTION:
Cellular senescence increases with aging and contributes to physiological dysfunction. Studies in animal models show that the flavonoid compound fisetin is an effective treatment for reducing cellular senescence and improving vascular function with aging. No published studies have used fisetin to target cellular senescence in older adults to improve vascular function. In addition, the biological reasons (mechanisms) by which fistin may improve vascular function in older adults has not been assessed. This study will evaluate if intermittent treatment with fisetin in older adults improves vascular function, reduces biological markers of cellular senescence, oxidative stress and inflammatory factors produced by senescent cells (i.e., senescence-associated secretory phenotype factors). The study will also evaluate safety, tolerability and adherence with fisetin treatment.

ELIGIBILITY:
Inclusion Criteria:

* Age 65 years or older
* Women must be postmenopausal
* Body mass index (BMI) <40 kg/m2
* Willing to accept random assignment
* Weight stable in the prior 2 months (<2 kg weight change) and willing to remain weight stable throughout the study
* Ability to understand study procedures and to comply with them for the entire length of the study
* No blood donation within 8 weeks prior to baseline testing; willingness to abstain from blood donation during the study and for 8 weeks after study completion
* Absence of established, serious, unstable, chronic clinical disease (e.g., unstable CVD) as determined by study physician of record based on subject medical history, physical examination, resting ECG and standard clinical blood chemistries

Exclusion Criteria:

* Inability to refrain from alcohol for 24 hours prior to outcome assessment
* Individuals taking fisetin, quercetin, luteolin, Dasatinib, piperlongumine or Navitoclax (supplements or drugs with established senolytic effects) within 6 months prior to baseline testing; should new research reveal other dietary supplements or drugs with potential senolytic effects, their use will be evaluated, and their use may lead to exclusion of the subject by the PI
* New use of regular cardiovascular-acting medication which, in the opinion of the PI, affects the outcomes of the study within 3 months prior to starting baseline testing as reported during medication review during screening (these individuals could be enrolled after 3 months of regular use)
* Chronic use of a dietary supplement which, in the opinion of the PI, affects the outcomes of the study, within 1 month prior to starting baseline testing as reported during medication review during screening (these individuals could be enrolled after 1 month of regular use)
* Active malignancy (including myeloma) or malignancy that was active within 5 years prior to baseline testing
* Inability or unwillingness of individual to give written informed consent
* Current or past participation within 3 months in another clinical trial that, in the opinion of the PI, would affect the outcomes of the study
* Known hypersensitivity or allergy to fisetin
* Blood donation within 2 months prior to baseline testing
* Resting blood pressure >160 mmHg systolic or >110 mmHg diastolic
* Regular vigorous aerobic/endurance exercise

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2023-09-25 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in endothelial function at 1 month | 1 month
  Brachial artery flow-mediated dilation

SECONDARY OUTCOMES:
Change from baseline in aortic stiffness at 1 month | 1 month
  Carotid-femoral pulse wave velocity

OTHER OUTCOMES:
Change from baseline in suppression of endothelial function by mitochondrial oxidative stress at 1 month | 1 month
  Change in brachial artery flow-mediated dilation with acute, supratherapeutic MitoQ (160mg)
Change from baseline in endothelial cell markers of cellular senescence at 1 month | 1 month
  Endothelial cell abundance of p16 and p21
Change from baseline in blood cell markers of cellular senescence at 1 month | 1 month
  p16-positive T-cells
Change from baseline in plasma markers of the senescence-associated secretory phenotype | 1 month
  Circulating pro-inflammatory cytokines and chemokines

CONTACTS AND LOCATIONS:
Overall Officials: Matthew J Rossman, PhD, Principal Investigator — University of Colorado, Boulder
Locations (1):
- University of Colorado Boulder, Boulder, Colorado, United States